CLINICAL TRIAL: NCT02670434
Title: Safety and Efficacy Comparison Study of NK-104-CR (Controled Release) in Patients With Primary Hyperlipidemia or Mixed Dyslipidemia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NK-104-CR-3.01US
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Hyperlipidemia; Dyslipidemia
MeSH Terms: conditions — Hyperlipidemias; Dyslipidemias | interventions — pitavastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- NK-104-CR (Experimental): Controlled release NK-104
  Interventions: Drug: NK-104-CR
- Placebo (Placebo Comparator): Livalo Placebo
  Interventions: Drug: Placebo
- Livalo® Immediate Release IR (Active Comparator): Immediate Release Livalo®
  Interventions: Drug: Livalo

INTERVENTIONS:
Drug: NK-104-CR — NK-104-CR 8 mg daily for 52 weeks
  Arms: NK-104-CR
Drug: Placebo — Placebo daily for 12 weeks
  Arms: Placebo
Drug: Livalo — Livalo® IR daily from week 12 to week 52
  Arms: Livalo® Immediate Release IR

SUMMARY:
The purpose of this study is to compare the efficacy of NK-104-CR with Placebo and Livalo® on the reduction of LDL-C and to evaluate the safety of NK-104-CR in patients with primary hyperlipidemia or mixed dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with primary hyperlipidemia or mixed dyslipidemia who are ≥18 and ≤80 years of age at the time of consent;
* Fasting plasma LDL-C ≥160 mg/dL and ≤250 mg/dL and TG values of ≤300 mg/dL
* Patients who are naïve to statin or who are able to safely discontinue the use of all lipid-lowering agents for 6 weeks before randomization and throughout study participation

Exclusion Criteria:

* Homozygous familial hypercholesterolemia;
* Any conditions which may cause secondary dyslipidemia.
* Newly diagnosed or poorly controlled diabetes mellitus as defined by HbA1c >8%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Percent change in LDL-C from baseline | 12 Weeks

SECONDARY OUTCOMES:
The percent change from baseline in fasting serum total cholesterol (TC ) | 12 Weeks

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Beverly Hills, California
  - Chino, California
  - Lincoln, California
  - Los Angeles, California
  - Newport Beach, California
  - North Hollywood, California
  - Thousand Oaks, California
  - Vista, California
  - Brooksville, Florida
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Port Orange, Florida
  - Marietta, Georgia
  - Meridian, Idaho
  - Chicago, Illinois
  - Evanston, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Newton, Kansas
  - Wichita, Kansas
  - Auburn, Maine
  - Elkridge, Maryland
  - Edina, Minnesota
  - Jackson, Mississippi
  - Butte, Montana
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Endwell, New York
  - Rochester, New York
  - Greensboro, North Carolina
  - Cincinnati, Ohio
  - Kettering, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Willoughby Hills, Ohio
  - Downingtown, Pennsylvania
  - Charleston, South Carolina
  - Mt. Pleasant, South Carolina
  - Kingsport, Tennessee
  - Houston, Texas
  - Hurst, Texas
  - Madison, Wisconsin